CLINICAL TRIAL: NCT05703971
Title: A Phase 1/2 Clinical Trial of Quaratusugene Ozeplasmid and Atezolizumab Maintenance Therapy in Patients With Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: Quaratusugene Ozeplasmid (Reqorsa) and Atezolizumab Maintenance Therapy in ES-SCLC Patients
Acronym: Acclaim-3
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genprex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONC-005
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: atezolizumab; atezolizumab and hyaluronidase-tqjs; Tumor Suppressor Gene 2 (TUSC2); Lipid Nanoparticle (LNP); Gene Therapy; TECENTRIQ; ES-SCLC; REQORSA; quaratusugene ozeplasmid
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1: 3+3 dose selection to identify RP2D. Phase 2: open label, non-randomized treatment with quaratusugene ozeplasmid at RP2D in combination with atezolizumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Up to 2 sequential dose selection cohorts will be treated with quaratusugene ozeplasmid (intravenous (IV) administration once every 21 days) plus atezolizumab (1200 mg IV administration once every 21 days) until disease progression or unacceptable toxicity.
  Quaratusugene ozeplasmid doses will be evaluated (0.09 [starting dose], and 0.12 mg/kg) until the RP2D is identified.
  Interventions: Biological: quaratusugene ozeplasmid; Biological: atezolizumab
- Phase 2 (Experimental): Patients will be treated with the RP2D of quaratusugene ozeplasmid (IV administration once every 21 days) plus atezolizumab (1200 mg IV administration once every 21 days) or atezolizumab and hyaluronidase-tqjs (15 mL subcutaneous [SQ] administration once every 21 days) until disease progression or unacceptable toxicity
  Interventions: Biological: quaratusugene ozeplasmid; Biological: atezolizumab

INTERVENTIONS:
Biological: quaratusugene ozeplasmid — Quaratusugene ozeplasmid is an experimental nonviral immunogene therapy utilizing the TUSC2 gene, designed to target cancer cells by interrupting cell signaling pathways that allow cancer cells to grow, reestablishing pathways that promote cancer cell death and modulating the immune response against cancer cells.
  Other Names: REQORSA
Biological: atezolizumab — Atezolizumab is a monoclonal antibody that belongs to a class of drugs that binds to the programmed death-receptor 1 ligand 1 (PD-L1), blocking the PD-1/PD-L1 pathway, thereby removing inhibition of the immune response, potentially breaking peripheral tolerance and inducing immune-mediated adverse reactions.
  Other Names: TECENTRIQ

SUMMARY:
This clinical trial will evaluate the combination of quaratusugene ozeplasmid with atezolizumab as maintenance therapy for patients with Extensive Stage Small Cell Lung Cancer (ES-SCLC).

The study is comprised of 2 phases, a dose selection phase (Phase 1) and a safety and efficacy evaluation phase (Phase 2).

DETAILED DESCRIPTION:
Acclaim-3 is an open-label, multi-center, Phase 1/2 study evaluating the combination of quaratusugene ozeplasmid with atezolizumab as maintenance therapy for patients with ES-SCLC who did not develop tumor progression after receiving at least 3 cycles, and no more than 4 cycles, of induction therapy with carboplatin plus etoposide and atezolizumab.

Toxicities will be assessed by the Investigator using United States National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Serious Adverse Events and Dose Limiting Toxicities (DLTs) will be reviewed by a safety review committee.

Phase 1: Enrollment in Phase 1 is complete and the recommended Phase 2 dose (RP2D) of quaratusugene ozeplasmid when given in combination with atezolizumab was determined.

Phase 2: Enrollment has been initiated and enrolled patients are treated with quaratusugene ozeplasmid at the RP2D in combination with atezolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years.
* Documented history of histologically or cytologically confirmed ES-SCLC, prior to starting treatment with the combination of atezolizumab, carboplatin, and etoposide
* Complete Response (CR), Partial Response (PR), or Stable Disease (SD) after receiving at least three cycles, and no more than four cycles, of atezolizumab, carboplatin, and etoposide.
* Eastern Cooperative Oncology Group performance status (ECOG PS) score from 0 to 1.
* Must be ≥28 days beyond major surgical procedures such as thoracotomy, laparotomy, or joint replacement, and must not have evidence of wound dehiscence, active wound infection, or comparable major residual complications of the surgery per Investigator assessment.
* Asymptomatic brain metastases must meet ALL criteria of the following (a-d):

  1. No history of seizures in the preceding six months.
  2. Definitive treatment must be completed ≥21 days prior to enrollment.
  3. Must be off steroids administered because of brain metastases or related symptoms for ≥7 days.
  4. If had previous brain irradiation, post-treatment imaging must demonstrate stability or regression of the brain metastases.
* Absolute neutrophil count (ANC) >1500/mm3, platelet count >100,000/mm3 within ≤28 days.
* Adequate renal function documented by serum creatinine of ≤1.5 mg/dL or calculated creatinine clearance >50 ml/min within ≤28 days.
* Adequate hepatic function as documented by serum bilirubin <1.5 mg/dL and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 X upper limit of normal (ULN) within ≤28 days.
* Stable cardiac condition with a left ventricular ejection fraction ≥40% within ≤28 days.
* If female of childbearing potential (FOCBP), must have negative serum pregnancy test (serum beta-human chorionic gonadotropin [β-hCG]) within ≤7 days of first dose.
* FOCBP and non-sterile men who are sexually active with FOCBP must agree to use two forms of contraception including one highly effective and one effective methods beginning ≥2 weeks prior to enrollment through for four months following the last dose of study treatment.
* If male, must agree to no sperm donation during study treatment and for an additional four months following the last dose of study treatment.
* Must have voluntarily signed an informed consent in accordance with institutional policies.

Exclusion Criteria:

* Unable to tolerate atezolizumab treatment, leading to early treatment discontinuation or prolonged/frequent dosage modifications in previous atezolizumab treatment as determined by the Investigator.
* Received prior gene therapy.
* Received prophylactic cranial irradiation or consolidation thoracic radiation.
* Active systemic viral, bacterial, or fungal infection(s) requiring treatment.
* Serious concurrent illness or psychological, familial, sociological, geographical, or other concomitant conditions that, in the opinion of the Investigator, would not permit adequate follow-up and compliance with the study protocol.
* History of autoimmune disease requiring immunosuppression.
* History of myocardial infarction or unstable angina within ≤6 months.
* Known human immunodeficiency virus (HIV) infection or has active hepatitis infection.
* Female who is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) - Phase 1 | First 21-days at each dose level
  The MTD and/or RP2D of the combination of quaratusugene ozeplasmid and atezolizumab.
  Note: if a MTD is not determined, the RP2D will be selected based on all available data (safety, PK, PD, and preliminary efficacy).
Progression-Free Survival Rate (PFSR) - Phase 2 | 18-weeks from Day 1 of maintenance therapy
  PFSR at 18 weeks according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Safety Profile - Phase 1 | Approximately 6 months
  Adverse events according to CTCAE v5.0
Progression-free Survival (PFS) - Phase 1 & Phase 2 | Approximately 5 months
  PFS per RECIST 1.1. PFS is defined as time from Day 1 of maintenance therapy to disease progression or death.
Pharmacokinetics (PK) of Quaratusugene Ozeplasmid - Phase 1 & Phase 2 | First 21-day treatment cycle
  Concentration of quaratusugene ozeplasmid in whole blood samples.
Overall Survival (OS) - Phase 1 & Phase 2 | Approximately 18 months
  Number of months from Day 1 of maintenance therapy to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Berger, MD, Study Director — Genprex, Inc.
Locations (13):
- United States (13):
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Gabrail Cancer Center Research, Canton, Ohio
  - Oncology_Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - Oncology_Hematology Care Clinical Trials, LLC, Fairfield, Ohio
  - Willamette Valley Cancer Institute (Oregon), Eugene, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Providence Cancer Institute, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - Texas Oncology - DFW, Dallas, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Northwest Cancer Specialists, P.C., Vancouver, Washington